CLINICAL TRIAL: NCT02792036
Title: Intravitreal Carboplatin for the Treatment of Participants With Recurrent or Refractory Intraocular Retinoblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: iRET; NCI-2016-00848 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2016-06-02; First posted 2016-06-07 (Estimated); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Retinoblastoma
MeSH Terms: conditions — Retinoblastoma | interventions — Carboplatin; Maxitrol; Anti-Infective Agents; Cryotherapy; Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Participants with retinoblastoma that is refractory or has relapsed inside the eye.
  Interventions: Carboplatin, Maxitrol® , focal therapy, plaque radiotherapy.
  Interventions: Drug: Carboplatin; Drug: Maxitrol®; Procedure: Focal Therapy; Procedure: Plaque Radiotherapy

INTERVENTIONS:
Drug: Carboplatin — Carboplatin will be given intravitreally. Participants are eligible to receive up to 8 injections per eye (once approximately every 14 days) based on lack of toxicity and evidence of tumor response. An injection of consolidation will be given once a complete response is observed. If further regression of "stable" seeds is noted, additional injections (up to 8 maximum per eye) will be provided at the discretion of the treating team. Injections could be repeated if vitreous recurrence occurs from another source (and patient has not reached 8 max limit per eye).
  Other Names: Paraplatin®
Drug: Maxitrol® — Maxitrol® contains neomycin and polymyxin B sulfates and dexamethasone ophthalmic suspension and is for topical ophthalmic use only. It will be given for continued use for five days following the carboplatin injection to prevent infection.
  Other Names: Anti-infective
Procedure: Focal Therapy — Simultaneously with intravitreal carboplatin, focal therapy will be applied as needed to eradicate the retinal source of the seeding as well as all epiretinal and subretinal active tumors at the discretion of the treating ocular oncologist.
  Other Names: Cryotherapy; Laser photocoagulation; Thermo-therapy
Procedure: Plaque Radiotherapy — Participants who have developed progressive disease despite focal (non-irradiative) therapy will receive brachytherapy determined by consensus between the treating ophthalmologist and radiation oncologist.
  Other Names: Brachytherapy

SUMMARY:
Retinoblastoma (RB) is the most common intraocular tumor of childhood. Recurrent or refractory disease following therapy most often occurs due to persistence of vitreous disease and/or retinal reactivation of the main tumor mass. With this treatment protocol, investigators seek to identify a less invasive method of local drug delivery that does not disrupt the eye's integrity.

PRIMARY OBJECTIVE:

* To determine the safety and toxicity profile associated with intravitreal carboplatin for the treatment of recurrent or progressive intraocular retinoblastoma with vitreous seeding.

SECONDARY OBJECTIVES:

* To estimate the ocular salvage rate after treatment with intravitreal carboplatin in patients with recurrent or progressive intraocular retinoblastoma with vitreous seeding.
* To evaluate the effects of intravitreal carboplatin therapy on the histopathology of eyes enucleated for progressive or recalcitrant disease while on therapy.

DETAILED DESCRIPTION:
The eye(s) will be sterilized prior to injection. Aqueous fluid (0.1-0.15ml) will be withdrawn and sent for pathology review. Carboplatin diluted in normal saline will be administered via intravitreal injection under anesthesia once to each eligible eye approximately every 14 days. Following the injection, triple freeze/thaw cryotherapy is applied to the injection site and the eye is washed with water. The eye is gently "shaken" in all directions to evenly distribute the drug.

This trial will use a traditional phase I design for dose de-escalation with two dose levels. The first 6 patients will be enrolled at dose level 1 and will be observed for dose-limiting toxicity (DLT) throughout the treatment period up to approximately 5 months after start of therapy. If 0-2 (of the first 6) participants experience DLT, a second cohort of 6 patients will be enrolled at the same dose level 1. Study accrual would be completed at 12.

However, if 3 or more of the first 6 patients experience DLT at dose level 1, the dose level would be de-escalated to level -1 and 6 patients enrolled at this level (dose -1). If 0-2 patients experience DLT at dose level -1, a second cohort of 6 patients will be enrolled at dose level -1, and the study accrual would be complete. If 3 or more patients experience DLT at dose level -1, accrual would also be complete.

ELIGIBILITY:
Inclusion Criteria:

* Refractory or recurrent retinoblastoma with vitreous seeding meeting eligibility criteria by ultrasonic biomicroscopy performed during examination under anesthesia (EUA) by an ophthalmologist:

  * At least three consecutive clock hours of disease-free, attached peripheral retina through which the intraocular injection may be administered.
  * Absence of invasion in anterior and posterior chamber.
  * Absence of anterior hyaloid detachment.
  * Absence of retinal detachment at the entry site.
  * Absence of tumor at the entry site.
* ECOG Performance Score must be ≤ 2 within two weeks prior to registration.
* Participants must have an adequate liver function, as defined by bilirubin ≤3 x upper limit of normal (ULN), and SGOT and SGPT ≤3 x ULN.
* Participants must have adequate renal function as defined by serum creatinine ≤3 x ULN for age.
* Legal guardians must sign an informed consent indicating that they are aware of this study, the possible benefits, and toxic side effects. Legal guardians will be given a signed copy of the consent form.

Exclusion Criteria:

* Presence of metastatic disease or gross orbital involvement.
* Participants must not have an invasive infection at time of protocol entry.
* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2019-10-04 (Actual); Study Completion 2019-10-04 (Actual)

PRIMARY OUTCOMES:
Number of participants who develop dose-limiting toxicity (DLT) | From baseline through end of therapy (up to 5 months)
  DLTs are defined as any of the following: uveitis, sterile or infectious endophthalmitis, retinopathy or rhegmatogenous retinal detachment, massive vitreous hemorrhage that obscures direct visualization of the retina/tumor, and/or cataract that threatens the visual axis or view by treating physician.
  Grade 3 or 4 allergic reactions should lead to discontinuation of intravitreal carboplatin injections. Patients who have grade 3 or 4 allergic reactions will not be evaluable for this objective and will be replaced.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Brennan, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols